CLINICAL TRIAL: NCT02832830
Title: Image-guided and Intensity-modulated Radiotherapy Versus External Beam Radiotherapy for Patients With Spine Metastases
Acronym: IRON-1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRON-1
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Vertebral Bony Metastases
Keywords: bony metastases; palliative radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): intensity modulated radiotherapy (IMRT) 10 x 3 Gy
  Interventions: Radiation: IMRT
- B (Active Comparator): fractionated conventional external beam RT 10×3 Gy
  Interventions: Radiation: fractionated RT

INTERVENTIONS:
Radiation: IMRT — Intensity modulated Raiotherapy (IMRT) of the involved spinal bone metastasis
  Arms: A
Radiation: fractionated RT — external beam Radiotherapy of the involved spinal bone metastasis
  Arms: B

SUMMARY:
The aim of this explorative trial is to verify the comparability of a fractionated intensity modulated radiotherapy with a conventional radiotherapy related to quality of life on the one hand and to evaluate toxicity, re-calcification and stability of vertebral body as well as pain relief and local response for palliative patients with painful spinal bone metastases on the other hand. This is a single-center, prospective randomized controlled trial with parallel-group design to determine the quality of life after RT in patients with spinal bone metastases. Two different techniques were evaluated: intensity modulated radiotherapy (IMRT) and fractionated conventional external beam RT with 10×3 Gy each.

Experimental intervention:

IMRT 10 x 3 Gy

Control intervention:

3D-RT 10 x 3 Gy

DETAILED DESCRIPTION:
The aim of this explorative trial is to verify the comparability of a fractionated intensity modulated radiotherapy with a conventional radiotherapy related to quality of life on the one hand and to evaluate toxicity, re-calcification and stability of vertebral body as well as pain relief and local response for palliative patients with painful spinal bone metastases on the other hand. This is a single-center, prospective randomized controlled trial with parallel-group design to determine the quality of life after RT in patients with spinal bone metastases. Two different techniques were evaluated: intensity modulated radiotherapy (IMRT) and fractionated conventional external beam RT with 10×3 Gy each.

Experimental intervention:

IMRT 10 x 3 Gy

Control intervention:

3D-RT 10 x 3 Gy After the baseline measurements have been recorded, the patients will be randomly assigned to one of the two groups: IMRT 10×3 Gy (n = 30) or fractionated conventional 3D-RT 10×3 Gy (n = 30). The RT will be applied daily (mondy to Friday).

Follow-up per patient:

The target parameters will be measured and recorded at baseline, at the end of RT (t1), and at 12 weeks (t2) and 6 months (t3) after the end of the irradiation period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically confirmed tumor diagnosis and with secondary diagnosed solitary/multiple spinal bone metastases
* Indication for RT of the spinal bone metastases
* Age of between 18 and 85 years
* Karnofsky index of at least 50
* Signed declaration of informed consent

Exclusion Criteria:

* Lymphoma
* Significant neurological or psychiatric disorders, including dementia and epileptic seizures
* Previous RT at the current irradiation site
* Other severe disorders that in the judgment of the study director may prevent the patient's participation in the study
* Lacking or diminished legal capacity
* Any medical of psychological condition that the study director considers a preventive factor for the patient's ability to complete the study or to adequately understand the scope of the study and to give his or her consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
quality of life | 3-months-time-point after the end of RT
  improvement of more than 10% according to the EORTC BM22 questionaire measured at the 3-months-time-point after the end of RT (t2).

SECONDARY OUTCOMES:
bone density | 12 weeks post completion radiotherapy
  bone density is assessed 12 weeks post completion of radiotherapy using follow-up CT scan of the spine
pain reduction | end of treatment, 12 and 24 weeks post completion of radiotherapy
  pain is evaluated using the VAS pain scale (0-100 points) at completion and 12/ 24 weeks post completion of radiation
Fatigue | 12 and 24 weeks post completion of therapy
  Fatigue is assessed using the EORTC FA13 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Radiation Oncology, University of Heidelberg, Germany, Heidelberg, Germany, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chung Y, Yoon HI, Kim JH, Nam KC, Koom WS. Is helical tomotherapy accurate and safe enough for spine stereotactic body radiotherapy? J Cancer Res Clin Oncol. 2013 Feb;139(2):243-8. doi: 10.1007/s00432-012-1321-0. Epub 2012 Oct 2. PMID 23052695
- [Result] Katsoulakis E, Riaz N, Cox B, Mechalakos J, Zatcky J, Bilsky M, Yamada Y. Delivering a third course of radiation to spine metastases using image-guided, intensity-modulated radiation therapy. J Neurosurg Spine. 2013 Jan;18(1):63-8. doi: 10.3171/2012.9.SPINE12433. Epub 2012 Oct 26. PMID 23101946
- [Result] Murai T, Murata R, Manabe Y, Sugie C, Tamura T, Ito H, Miyoshi Y, Shibamoto Y. Intensity modulated stereotactic body radiation therapy for single or multiple vertebral metastases with spinal cord compression. Pract Radiat Oncol. 2014 Nov-Dec;4(6):e231-7. doi: 10.1016/j.prro.2014.02.005. Epub 2014 Mar 31. PMID 25407874
- [Result] Wu JS, Wong R, Johnston M, Bezjak A, Whelan T; Cancer Care Ontario Practice Guidelines Initiative Supportive Care Group. Meta-analysis of dose-fractionation radiotherapy trials for the palliation of painful bone metastases. Int J Radiat Oncol Biol Phys. 2003 Mar 1;55(3):594-605. doi: 10.1016/s0360-3016(02)04147-0. PMID 12573746
- [Derived] Sprave T, Verma V, Forster R, Schlampp I, Hees K, Bruckner T, Bostel T, El Shafie RA, Welzel T, Nicolay NH, Debus J, Rief H. Bone density and pain response following intensity-modulated radiotherapy versus three-dimensional conformal radiotherapy for vertebral metastases - secondary results of a randomized trial. Radiat Oncol. 2018 Oct 30;13(1):212. doi: 10.1186/s13014-018-1161-4. PMID 30376859
- [Derived] Meyerhof E, Sprave T, Welte SE, Nicolay NH, Forster R, Bostel T, Bruckner T, Schlampp I, Debus J, Rief H. Radiation-induced toxicity after image-guided and intensity-modulated radiotherapy versus external beam radiotherapy for patients with spinal bone metastases (IRON-1): a study protocol for a randomized controlled pilot trial. Trials. 2017 Mar 3;18(1):98. doi: 10.1186/s13063-017-1847-1. PMID 28253920